CLINICAL TRIAL: NCT01478568
Title: An Open-label, One-sequence Crossover Study to Evaluate the Effect of Multiple Doses of YM178 on the Pharmacokinetics of the CYP2D6 Substrate Desipramine in Healthy Subjects
Brief Title: To Evaluate the Effect of Mirabegron (YM178) on Blood Levels of Desipramine When They Are Taken Together
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None
Other Study IDs: 178-CL-058; 2008-000215-15 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2013-07

CONDITIONS: Pharmacokinetics of Mirabegron; Healthy Subjects
Keywords: Pharmacokinetics; Mirabegron; Phase 1
MeSH Terms: interventions — mirabegron; Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mirabegron / desipramine (Experimental)
  Interventions: Drug: mirabegron; Drug: desipramine

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178
Drug: desipramine — oral
  Other Names: pertofrane; norpramin

SUMMARY:
The study aims to evaluate if blood levels of desipramine change whilst being dosed at the same time with daily mirabegron.

DETAILED DESCRIPTION:
This is an open-label, one-sequence crossover design study to evaluate the drug-drug interaction between mirabegron and desipramine. The effect of mirabegron on the plasma concentration of desipramine will be evaluated after 13 day repeated administration. The recovery of CYP2D6 activity is also being explored by comparing the pharmacokinetic profiles of desipramine after a 2 week wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18.5 and 30.0 kg/m2 inclusive
* Subject is genotyped and phenotyped as an extensive metabolizer for CYP2D6

Exclusion Criteria:

* Known or suspected hypersensitivity to YM178 or any of the components of the formulation used
* Known or suspected hypersensitivity to desipramine or any of the components of the formulation used
* Pregnant or breast feeding within 6 months before screening assessment
* Any clinical history of major depressive disorder, cardiovascular disease, urinary retention, glaucoma, thyroid disease and/or seizure disorder
* Any of the liver function tests (i.e. Alanine Aminotransferase (ALT), Asparate Aminotransferase (AST) and Alkaline phosphatase) above the upper limit of normal at repeated measurements
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug (excluding non-active hay fever)
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* Abnormal pulse rate and/or blood pressure measurements at the pre-study visit as follows: pulse rate <40 or >90 bpm; mean systolic blood pressure >140 mmHg; mean diastolic blood pressure >90 mmHg (blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse rate will be measured automatically)
* A marked baseline prolongation of QT/QTc interval after repeated measurements of >450 ms, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of desipramine assessed by plasma concentration while at steady state levels of mirabegron | Pre-dose until 72 hours after dosing

SECONDARY OUTCOMES:
Monitoring of safety and tolerability through assessment of vital signs, ECG, clinical safety laboratory and adverse events | Baseline until End of Study Visit (7 to 14 days after last dose)
Pharmacokinetics of desipramine assessed by plasma concentration after wash-out of mirabegron | Pre-dose until 72 hours after wash-out

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- SGS Aster, Paris, France

REFERENCES:
- [Background] Krauwinkel W, Dickinson J, Schaddelee M, Meijer J, Tretter R, van de Wetering J, Strabach G, van Gelderen M. The effect of mirabegron, a potent and selective beta3-adrenoceptor agonist, on the pharmacokinetics of CYP2D6 substrates desipramine and metoprolol. Eur J Drug Metab Pharmacokinet. 2014 Mar;39(1):43-52. doi: 10.1007/s13318-013-0133-1. Epub 2013 Jun 1. PMID 23728524